CLINICAL TRIAL: NCT06255041
Title: A Double-Blind Observational Study to Evaluate the Ability of Trained Detection Dogs to Detect Cancer in Breath Samples: The Rainbow Study
Brief Title: Detection of Cancer in Breath Samples by Trained Detection Dogs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SpotitEarly (Industry)
Responsible Party: Sponsor
Other Study IDs: SIE-001
Record Dates: First submitted 2024-02-04; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Colorectal Cancer; PROSTATE CANCER; Lung Cancer
Keywords: Breath Sample; Detection Dogs; Cancer Screening
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to show that trained detection dogs can identify breast, lung, prostate or colorectal cancer by sniffing masks containing breath samples. In this study, individuals who will undergo cancer screening at an integrated cancer prevention center or biopsy for a suspected malignancy, will be asked to provide a breath sample by breathing into a surgical mask. The mask will then be sent to the laboratory, where trained detection dogs will determine if the person who provided the mask has breast, lung, prostate or colorectal cancer or if the person does not have these types of cancer. The results provided by the dogs will be compared to the actual cancer screening results or biopsy results in order to determine the accuracy of cancer detection by the trained dogs.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 and over.
2. Signing an informed consent prior to performing the test.
3. Intended to undergo screening tests for cancer detection.
4. Did not smoke 2 hours before providing the breath sample
5. Did not drink coffee in the hour before providing the breath sample
6. Did not drink an alcoholic beverage in the hour prior to providing the breath sample.
7. Did not eat food in the hour before providing the breath sample.

Exclusion Criteria:

1. Was diagnosed with cancer or was treated for cancer in the seven years preceding the study, excluding non-metastatic skin tumors that were surgically removed.
2. Undergoing chemotherapy for any purpose.
3. Pregnant or breastfeeding
4. Had a medical procedure in the chest cavity and/or airways in the two weeks prior to providing the breath sample that may interfere with the ability to correctly provide a breath sample.
5. Has a Helicobacter pylori infection.
6. Has a peptic ulcer disease.
7. Has a flare-up of an inflammatory bowel disease (Crohn's disease/ulcerative colitis).
8. has an active infection, such as COVID-19, abscess, bacterial/viral/fungal infection, pneumonia, laryngitis, intestinal inflammation, active tuberculosis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women over the age of 18 undergoing screening for early detection of breast cancer, colon cancer, lung cancer, and prostate cancer at the medical centers participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Specificity of detection of any cancer (breast, lung, prostate or colorectal cancer) by the breath test. | 2 years
  Specificity is defined as the number of participants who were identified by the breath sample test as negative for cancer divided by the number of participants who were identified by the gold standard test as being negative for cancer.
Sensitivity of detection of any cancer (breast, lung, prostate or colorectal cancer) by the breath test. | 2 years
  Sensitivity is defined as the number of participants who were identified by the breath sample test as positive for cancer divided by the number of participants who were identified by the gold standard test as being positive for cancer.

SECONDARY OUTCOMES:
Specificity, sensitivity, negative predictive value, and positive predictive value of the breath test for detecting breast cancer | 2 years
Specificity, sensitivity, negative predictive value, and positive predictive value of the breath test for detecting colorectal cancer | 2 years
Specificity, sensitivity, negative predictive value, and positive predictive value of the breath test for detecting lung cancer | 2 years
Specificity, sensitivity, negative predictive value, and positive predictive value of the breath test for detecting prostate cancer | 2 years
The rate of early-stage cancer cases detected by the breath test | 2 years
Inter-observer variability among the detection dogs | 2 years
Intra-observer variability among the detection dogs | 2 years

OTHER OUTCOMES:
The detection rate of types of cancer that the dog was not trained to detect | 2 years
The rate of cancer detection among participants identified as negative by biopsy and positive by the breath test | 2 years
The duration for which a breath sample remains effective for detection by a detection dog | 2 years
The duration for which a breath sample collected on an alternative mask substrate remains effective for detection by a detection dog | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Arber, Principal Investigator — Tel-Aviv Sourasky Medical Center; Elizabeth Half, Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No